CLINICAL TRIAL: NCT00574782
Title: Evaluation of the Efficacy of Rosuvastatin in Daily Practice in Untreated High Risk Patients (CHALLENGE)
Acronym: CHALLENGE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NL950057
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease; Peripheral Vascular Disease; CVA; Diabetes
Keywords: cholesterol, coronary heart disease; rosuvastatin; LDL-C goal; hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease; Peripheral Vascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
In an observational multi-centre study (CHALLENGE), the effects were assessed of starting treatment with low doses of rosuvastatin in statin naive patients with a history of coronary heart disease (CHD), peripheral vascular disease (PVD), cerebrovascular accident (CVA), transient ischemic attack (TIA) or diabetes (DM), on low-density lipoprotein cholesterol (LDL-C) goal achievement. Also proportional changes in LDL-C, high-density lipoprotein cholesterol (HDL-C), total cholesterol (TC), triglycerides (TG) and the ratio TC/HDL-C were studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the study were high-risk patients with a documented history of CHD, PVD, cerebrovascular atherosclerotic disease, DM II or DM I with microalbuminuria. LDL-C had to be > 2.5 mmol/l and the patient did not use any cholesterol lowering medication during the last 3 months preceding inclusion. The specialist made the decision to start treatment with rosuvastatin irrespective of study participation. Patient approved to place anonymous results at the disposal of AstraZeneca

Exclusion Criteria:

* Exclusion criteria included patients familiar with muscular pain, myopathy or liver function disorders (inclusive elevation of serum transaminases), patients with familial dyslipideamia like familial hypercholesterolaemia and familial combined hyperlipid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2660 (Actual)
Dates: Start 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid van Geel, Study Chair — CV; Ingeborg Vosjan, Study Chair — CV